CLINICAL TRIAL: NCT06055920
Title: PEERLESS II: RCT of FlowTriever vs. Anticoagulation Alone in Pulmonary Embolism
Brief Title: The PEERLESS II Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-001
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Anticoagulants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FlowTriever (Active Comparator): Mechanical thrombectomy for pulmonary embolism using the FlowTriever System.
  Interventions: Device: FlowTriever System
- Anticoagulation (Active Comparator): Commercially available/market approved anticoagulation medication including but not limited to: Heparin Sodium, Coumadin, Rivaroxaban, Apixaban, etc.
  Anticoagulants are a group of medications that decrease your blood's ability to clot.
  Interventions: Drug: Anticoagulation Agents

INTERVENTIONS:
Device: FlowTriever System — Mechanical Thrombectomy for pulmonary embolism
  Arms: FlowTriever
Drug: Anticoagulation Agents — Commercially available/market approved anticoagulation medication including but not limited to: Heparin Sodium, Coumadin, Rivaroxaban, Apixaban, etc.
  Anticoagulants are a group of medications that decrease your blood's ability to clot.
  Arms: Anticoagulation

SUMMARY:
This study is a prospective, multicenter, randomized controlled trial of the FlowTriever System plus anticoagulation compared to anticoagulation alone for intermediate-risk acute PE.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment ≥ 18 years
2. Objective evidence of a proximal filling defect in at least one main or lobar pulmonary artery, as confirmed by CTPA, pulmonary angiography, or other imaging modality
3. RV dysfunction, as defined as one or more of the following: RV/LV ratio ≥ 0.9 or RV dilation or hypokinesis
4. At least two additional risk factors, identified by at least one measure in two separate categories noted below:

   a. Hemodynamic: i. SBP 90-100mmHg ii. Resting heart rate > 100 bpm b. Biomarker: i. Elevated* cardiac troponin (troponin I or troponin T, conventional or high sensitivity) ii. Elevated* BNP or NT-proBNP iii. Elevated venous lactate ≥2 mmol/L * Elevated, meaning at or above the upper limit of normal, per local standards for the assay used c. Respiratory: i. O2 saturation < 90% on room air ii. Supplemental O2 requirement ≥ 4 L/min iii. Respiratory rate ≥ 20 breaths/min iv. mMRC score > 0
5. Symptom onset within 14 days of confirmed PE diagnosis
6. Willing and able to provide informed consent

Exclusion Criteria:

1. Unable to be anticoagulated with heparin, enoxaparin or other parenteral antithrombin
2. Presentation with hemodynamic instability* that meets the high-risk PE definition in the 2019 ESC Guidelines1, including ANY of the following

   1. Cardiac arrest OR
   2. Systolic BP < 90 mmHg or vasopressors required to achieve a BP ≥ 90 mmHg despite adequate filling status, AND end-organ hypoperfusion OR
   3. Systolic BP < 90 mmHg or systolic BP drop ≥ 40 mmHg, lasting longer than 15 min and not caused by new-onset arrhythmia, hypovolemia, or sepsis * Patients who are stable at time of screening or randomization (i.e., SBP ≥ 90 mmHg and adequate organ perfusion without catecholamine or vasopressor infusion) may be included despite initial presentation including temporary, low-dose catecholamines or vasopressors, or temporary fluid resuscitation.
3. Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated
4. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the patient is not appropriate for catheter-based intervention (e.g., inability to navigate to target location, clot limited to segmental/subsegmental distribution, predominately chronic clot)
5. End stage medical condition with life expectancy < 3 months, as determined by the Investigator
6. Current participation in another drug or device study that, in the investigator's opinion, would interfere with participation in this study
7. Current or history of chronic thromboembolic pulmonary hypertension (CTEPH) or chronic thromboembolic disease (CTED) diagnosis, per 2019 ESC Guidelines1
8. If objective testing was performed*, estimated RV systolic pressure > 70 mmHg on standard of care echocardiography * If clinical suspicion of acute-on-chronic PE, chronic obstruction, or chronic thromboembolism, echocardiographic estimated RVSP must be confirmed ≤70 mmHg to meet eligibility. Pressure assessment not required if Investigator attests to absence of such clinical suspicion
9. Administration of advanced therapies (thrombolytic bolus, thrombolytic drip/infusion, catheter-directed thrombolytic therapy, mechanical thrombectomy, or ECMO) for the index PE event within 30 days prior to enrollment
10. Ventricular arrhythmias refractory to treatment at the time of enrollment
11. Known to have heparin-induced thrombocytopenia (HIT)
12. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being or that could prevent, limit, or confound the protocol-specified assessments). This includes a contraindication to use of FlowTriever System per local approved labeling
13. Subject is currently pregnant
14. Subject has previously completed or withdrawn from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Composite clinical endpoint constructed as a win ratio, a hierarchy of the following, which are assessed post-randomization: | through discharge or 30 days, whichever is sooner / dyspnea at 48 hours
  * All-cause mortality by 30 days, or
  * Clinical deterioration, defined by hemodynamic or respiratory worsening, through discharge or up to 30 days after randomization, whichever is sooner, or
  * All-cause hospital re-admission by 30 days, or
  * Bailout therapy, either after a deterioration or after documented failure to progress, through discharge or up to 30 days after randomization, whichever is sooner, or
  * Change in Dyspnea, by mMRC from Baseline to the 48-hour visit

SECONDARY OUTCOMES:
Composite clinical endpoint constructed as a win ratio hierarchy of the following three components, assessed post randomization: | up to 30 days
  * All-cause mortality, by 30 days, or
  * Clinical deterioration defined by hemodynamic or respiratory worsening, through discharge or up to 30 days after randomization, whichever is sooner, or
  * All-cause readmission, by 30 days
All-cause and PE-related mortality | At 30 and 90 days
All-cause and PE-related readmissions | At 30 and 90 days
Clinical deterioration | Through discharge or up to 30 days after randomization, whichever is sooner
  defined by hemodynamic or respiratory worsening
Bailout therapy | Through discharge or up to 30 days after randomization, whichever is sooner
  either after a deterioration or after documented failure to progress,
Major Bleeding, defined by the Bleeding Academic Research Consortium (BARC), level 3b, 3c, 5a, or 5b | At 30 and 90 days
  3b: Overt bleeding plus hemoglobin drop of ≥ 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade, bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid); bleeding requiring intravenous vasoactive agents 3c: Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal), subcategories confirmed by autopsy or imaging or lumbar puncture, intraocular bleed compromising vision.
  5a: Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious 5b: Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation
Dyspnea severity by mMRC score | At the 48-hour, 1-month, and 3-month visits
  0, no breathlessness except on strenuous exercise;
  * 1, shortness of breath when hurrying on the level or walking up a slight hill;
  * 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level;
  * 3, stops for breath after walking ∼100 m or after few minutes on the level; and
  * 4, too breathless to leave the house, or breathless when dressing or undressing
PE-related quality of life, by PEmb-QoL | At the 1- and 3-month visits
  Pulmonary Embolism Quality of Life: (higher = better)
General health-related quality of life, by EQ-5D-5L | At the 1- and 3-month visits
  Higher score = worse
6-minute walk distance | At the 1-month visit
RV/LV ratio | At the 48-hour visit
Post-PE Impairment diagnosis (PPEI) | Through the 3-month visit

CONTACTS AND LOCATIONS:
Overall Officials: Frances Mae West, MD, Principal Investigator — Jefferson Health; Jay Giri, MD, Principal Investigator — Penn Medicine; Bernhard Gebauer, MD, Principal Investigator — Charité University Hospital Berlin; Felix Mahfoud, MD, Principal Investigator — Universitaetsspital Basel
Locations (83):
- United States (50):
  - UAB Division of Cardiovascular Disease, Birmingham, Alabama
  - Brookwood Medical Center, Birmingham, Alabama
  - Huntington Memorial Hospital, Pasadena, California
  - University of Colorado, Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - HCA FL Largo Medical Center, Largo, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Baptist Health Louisville, Louisville, Kentucky
  - McLaren Greater Lansing, Lansing, Michigan
  - Metropolitan Heart & Vascular Institute, Coon Rapids, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Virtua Health, Camden, New Jersey
  - Valley Health, Ridgewood, New Jersey
  - SUNY, The University of Buffalo/Gates Vascular, Buffalo, New York
  - Northwell Health, New York, New York
  - Jamaica Hospital, Queens, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University - Wexner Medical Center, Columbus, Ohio
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - AHN Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - Wellspan York Hospital, York, Pennsylvania
  - HCA Tristar, Brentwood, Tennessee
  - UTMC Knoxville, Knoxville, Tennessee
  - Ascension Saint Thomas Hospital, Nashville, Tennessee
  - Parkland Hospital, Dallas, Texas
  - Texas Health Harris Methodist Hospital, Fort Worth, Texas
  - Methodist Main Hospital, San Antonio, Texas
  - Baylor Scott & White - Temple, Temple, Texas
  - Inova Fairfax, Falls Church, Virginia
  - Sentara Vascular Specialists, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - West Virginia University Ruby Memorial Hospital, Morgantown, West Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Onze Lieve Vrouwziekenhuis, Aalst, Belgium
- Canada (3):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
- Aarhus University Hospital, Aarhus, Denmark
- France (4):
  - CHU Lille, Lille
  - Hôpital Louis Pradel, Lyon
  - AP-HM Hopital La Timone, Marseille
  - Hôpital Nord Marseille, Marseille
- Germany (19):
  - University Hospital Augsburg, Augsburg
  - Universitäts-Herzzentrum Bad Krozingen, Bad Krozingen
  - Charité Campus Virchow Clinic - Klinik fuer Radiologie, Berlin
  - Unfall Krankenhaus Berlin, Berlin
  - University Hospital Cologne, Cologne
  - HerzZentrum Dresden Universitaetsklinik, Dresden
  - Universitaetsklinikum Dὒsseldorf, Düsseldorf
  - Elisabeth Hospital GmbH, Essen
  - Universitaetsklinikum Essen, Essen
  - CCB Frankfurt, Frankfurt
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - University Hospital - Heidelberg, Heidelberg
  - Universitaetsklinikum Saarlandes Homburg, Homburg
  - Westpfalz Klinikum, Kaiserslautern
  - Klinikum rechts der Isar (TUM), Munich
  - Ludwig Maximilians-University, Munich
  - University Hospital Regensburg, Regensburg
  - Helios Kliniken Schwerin, Schwerin
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen
- John Paul II Hospital, Krakow, Poland
- Hopital Clinico Universitario San Carlos, Madrid, Spain
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Universitätsspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giri J, Mahfoud F, Gebauer B, Andersen A, Friedman O, Gandhi RT, Jaber WA, Pereira K, West FM. PEERLESS II: A Randomized Controlled Trial of Large-Bore Thrombectomy Versus Anticoagulation in Intermediate-Risk Pulmonary Embolism. J Soc Cardiovasc Angiogr Interv. 2024 May 3;3(6):101982. doi: 10.1016/j.jscai.2024.101982. eCollection 2024 Jun. PMID 39132600